CLINICAL TRIAL: NCT02443259
Title: Short Term Neurobehavioural Outcomes in Late Preterm Neonates Born to Pre Eclamptic Mothers : a Prospective Observational Study
Brief Title: Neurobehavioural Outcomes in Late Preterm Neonates
Acronym: PRENB
Status: Completed | Type: Observational
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, DR VIKRAM DATTA, Lady Hardinge Medical College
Other Study IDs: LHMC/ECHR/2014/165
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Pre-Eclampsia
Keywords: NAPI; late preterm
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- late preterms from pre eclamptic mothers: late preterms born to pre eclamptic mothers
- late preterms: late preterm neonates

SUMMARY:
Hypertensive disorders are the most common medical complications in pregnancy and major causes of maternal, fetal, and neonatal morbidity and mortality. Fifty percent of hypertensive disorders of pregnancy are defined as pre eclampsia, the most important manifestation of the disease.

Preeclampsia is also a significant risk factor in the development of IUGR and represents the most common cause of IUGR in the nonanomalous infant. The incidence of thrombocytopenia, neutropenia and Bronchopulmonary dysplasia is also increased in neonates with preeclampsia.

The neurodevelopmental outcomes infants exposed to preeclampsia are highly variable. The study by Gray et al showed that preeclampsia is associated with a decreased risk of cerebral palsy. They also found a protective effect of maternal preeclampsia on cerebral palsy regardless of exposure to magnesium sulfate. However, contrary to this, study conducted by Shao-Wen Cheng et al has showed that infants born to pre-eclamptic mothers had lower MDI scores at 24 months of age (P= 0.04) as compared to infants without maternal pre-eclampsia. The study by Szymonowicz et al showed that neonates born to pre-eclamptic mothers had a significantly lower mean mental developmental index, and significantly more of these children had one or more impairments compared with the control group at 2 years of age. The neurodevelopmental outcomes in neonates born to preeclamptic mothers therefore remain inconclusive. Recently the role of neurobehaviour being evaluated early at 37-40 weeks of CGA is being predicted as an useful adjunct to the 12-18 month full neurodevelopmental assessment. This assumes significance in the context of initiation of early stimulation and objectivised individual developmental rehabilitation regimens for these infants.

DETAILED DESCRIPTION:
Preeclampsia is a multiorgan, heterogeneous disorder of pregnancy associated with significant maternal and neonatal morbidity and mortality.

The incidence of preeclampsia is about 5% to 10% of all pregnancies, with higher rates reported in first pregnancies, twin pregnancies, and in women who have had previous pre eclampsia. Fifty percent of hypertensive disorders of pregnancy are defined as preeclampsia, the most important manifestation of the disease.

While preeclampsia complicates 6%-10% of all pregnancies in the United States, the incidence is believed to be even higher in underdeveloped countries.

Perinatal mortality rates from range from 59 in 1,000 in developed countries to more than 300 in 1,000 in low income countries.

Preeclampsia and eclampsia accounts for 24% of all maternal deaths in india. Diagnostic criteria for preeclampsia Blood pressure Greater than or equal to 140 mm hg systolic or greater than or equal to 90 mm hg diastolic on two occasions at least 4 hours apart after 20 weeks of gestation in a woman with previously normal blood pressure Greater than or equal to 160 mm hg systolic or greater than or equal to 110 mm hg diastolic , hypertension can be confirmed within a short interval ( minutes ) to facilitate timely antihypertensive therapy And Proteinuria Greater than or equal to 300 mg per 24 hour urine collection ( or this amount extrapolated from a timed collection ) or Protein / creatinine ratio greater than or equal to 0.3 mg/dl Dipstick reading of 1+( used only if other quantitative methods not available )

Or in the absence of proteinuria, new onset hypertension with the new onset of any of the following:

Thrombocytopenia Platelet count less than 100000/ microliter Renal insufficiency Serum creatinine concentrations greater than 1.1 mg/dl or a doubling of the serum creatinine concentration in the absence of other renal disease Impaired liver function Elevated blood concentrations of liver transaminases to twice normal concentration Pulmonary edema Cerebral or visual symptoms

LATE PRETERMS: A SPECIAL COHORT

Definition:

Premature infants ( born at < 37 completed weeks gestation) are categorized into subgroups

* Very preterm (<32 completed weeks)
* Moderately preterm (between 32 and 33 completed weeks)
* Late preterm (between 34 and 36 completed weeks) Late preterm birth is an accepted term used for infants born at 34 0/7 to 36 +6/7 weeks gestation. This group was initially referred to as near term, but misleading implications of maturity has prompted the name change to late preterm.

Magnitude of late preterm births Prematurity is a leading cause of morbidity and mortality globally. Advances in medicine and technology have shifted the distribution of births away from term/post-term towards earlier gestations.

The percentage of live births in the United States that were born late preterm increased between 1990 and 2006 from 7.3% to 9.14% , a 25% increase.

This increase accounted for 84% of the increase in the prematurity during that same 16 year period. Thus this group of late preterms account for the maximum burden of premature births.

Etiology of late preterm births Preterm deliveries are divided into two groups

* The first group: Spontaneous late preterm births (premature labor with intact membranes or premature rupture of membranes) where there is limited control on preventing the birth and the focus lies in a better understanding of the management of the neonate in the perinatal period.
* The second group includes premature babies born after the induction of labor or performance of a cesarean section for maternal or fetal indications.

Consequences of late preterm births Acute Medical Morbidities and Mortality

This group is characterized by physiological immaturity with limited compensatory responses to extrauterine environment compared to term infants. They have greater risk than term babies for morbidities and mortalities such as:

* Temperature instability
* Hypoglycemia
* Respiratory distress
* Apnea
* Jaundice
* Feeding difficulties
* Dehydration
* Suspected sepsis
* Neurologic disorder and/or death The risk of death and/or a severe neurologic disorder defined by ischemic encephalopathy,Grade 3 or 4 IVH, cystic periventricular leukomalacia and/or seizures increased to 1.7% at 34 Weeks gestation as compared to 0.15% at 38 weeks gestation.

Long-term morbidities in late preterms Long-term outcomes affected by late preterm involve school performance, behaviour problems, social and medical disabilities, and mortality. Although the absolute risk of poor long-term outcomes in infants born late preterm are small, the risks are significantly greater than if born at 39-40 week gestation.Medical and social morbidities increase with decreasing gestational age. In cohort of 903,402 Norwegian infants born alive without congenital anomalies and followed through early adulthood, infants born late preterm had significant higher risks for cerebral palsy; cognitive dysfunction; schizophrenia; disorders of psychological development, behavior, and other major disabilities.

EFFECTS OF PREECLAMPSIA ON LATE-PRETERM INFANT OUTCOMES Risk of Fetal Demise/Stillbirth Severe preeclampsia represents significant risk factor for intrauterine fetal demise, with estimated stillbirth rate of 21 per 1000 20. In the setting of severe preeclampsia, the risk of fetal death outweighs the potential benefits of pregnancy prolongation. However, in cases of mild preeclampsia, the risk of fetal demise is over 50% less than pregnancies with severe preeclampsia (stillbirth rate of 9 per 1000) Intrauterine Growth Restriction (IUGR) Preeclampsia, a condition characterized by decreased uteroplacental blood flow and ischemia, is a significant risk factor in the development of IUGR and represents the most common cause of IUGR in the nonanomalous infant.

Hematologic Effects Maternal preeclampsia can result in neonatal thrombocytopenia, typically defined as a platelet count less than 150,000/uL. Severity of thrombocytopenia related to preeclampsia is highly variable, with a small percentage of infants developing severe or clinically significant thrombocytopenia (<50,000/uL). In addition to the well-described effects of preeclampsia on platelets, neonates delivered to women with preeclampsia have a 50% incidence of neutropenia (defined as absolute neutrophil count less than 500).

Bronchopulmonary Dysplasia (BPD) The study by Hansen et al shows that maternal preeclampsia is, associated with an increased risk for development of BPD, even after adjusting for gestational age, birth weight, and other clinical confounders (OR 2.96, 95% CI 1.17-7.51)

ELIGIBILITY:
INCLUSION CRITERIA

* Late preterm infants
* Pre eclampsia in mothers
* Parental Consent

EXCLUSION CRITERIA

* Major congenital malformation
* Eclampsia ( seizures in mother)
* Mothers on antipsychotic drugs
* Clinical Chorioamnionitis ( fever > 100.4º F, uterine fundal tenderness, maternal tachycardia (>100/min), fetal tachycardia (>160/min) and purulent or foul amniotic fluid )
* Birth Asphyxia (Apgar score of less than 7 at 1 minute of age)
* Multiple gestation.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: SAMPLE SIZE 60 intramural neonates divided in a group of 30 each. STUDY SUBJECTS Thirty late-preterm infants born to mothers with preeclampsia ---late preterms defined as infants born between 34 0/7 weeks and 36 6/7 weeks of gestation.
  CONTROL SUBJECTS Thirty late preterm infants born to mothers without preeclampsia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral score by NAPI at 40 weeks of corrected gestation for MDV(Motor development- vigor) and AO(Alertness-orientation) | 22 MONTHS
  Neurobehavioral score by NAPI at 40 weeks of corrected gestation for MDV(Motor development- vigor) and AO(Alertness-orientation)

SECONDARY OUTCOMES:
Incidence of small for gestational age babies. | 22 MONTHS
  Incidence of small for gestational age babies.
Need for NICU admission | 22 MONTHS
  Need for NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: vikram da datta, MD, Principal Investigator — LHMC
Locations (1):
- Lady Hardinge Medical College,New Delhi, Delhi, India